CLINICAL TRIAL: NCT03548740
Title: Diversity Analysis of Vaginal Microbiota on Women With High-risk Human Papillomavirus Infection and Cervical Cytological Abnormalities.
Brief Title: Diversity Analysis of Vaginal Microbiota on Women With High-risk Human Papillomavirus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, shuwang, Associate Professor, Peking Union Medical College Hospital
Other Study IDs: WS-1
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A
  Interventions: Biological: Human Papillomavirus
- Group B

INTERVENTIONS:
Biological: Human Papillomavirus — women with high-risk Human Papillomavirus or not
  Groups: Group A

SUMMARY:
Since other genital infections enhance HIV susceptibility by inducing inflammation, the investigators study the relationship between the vaginal microbiota composition and the risk of HPV infection, cervical cytological abnormalities.

DETAILED DESCRIPTION:
Persistent infection with oncogenic Human Papillomavirus (HPV) is necessary but not sufficient for the development of cervical cancer. Additional factors correlated with HPV persistence include immunodeficiency caused by HIV, smoking, use of oral contraceptives and, more recently reported, vaginal dysbiosis. In a state of dysbiosis, there is a marked reduction of Lactobacillus and a high diversity of bacteria, with increased abundance of anaerobic bacterial species. Based on this, the investigators are going to analyze the changes of microbiota in women with high-risk HPV and the cervical lesions. And the investigators hope to figure out the difference and change in microbiota to realize the tanning of cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of HR-HPV results.

Exclusion Criteria:

Clinical diagnosis of vaginitis, immune disease, malignancy History of cervical lesions Pregnancy Clinical diagnosis of other serious systemic primary diseases, such as severe liver and kidney dysfunction Severe mental illness

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group A: HPV positive, and the participants who have not taken drugs and physical therapy in the past six months, nor have chronic diseases (such as DM), take their vaginal microorganisms (do not mention the past History issues). Group B: HPV negative in the past 12 months, taking the vaginal microorganisms.
Sampling Method: Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Vaginal microbiota and HR-HPV infection | 12 months
  The persistence vaginal organism in HPV infection participants
Vaginal microbiota and the cervical lesion | 12 to 36 months
  The cervical cytology, HPV and the vaginal microbiota were evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China